CLINICAL TRIAL: NCT07251829
Title: Neoadjuvant Embolization and Cytoreduction to Ameliorate Radiotherapy Toxicity in Prostate Cancer
Brief Title: Neoadjuvant Embolization and Cytoreduction in Prostate Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Srinivas Raman (Other)
Responsible Party: Sponsor-Investigator, Srinivas Raman, MD, FRCPC, British Columbia Cancer Agency
Organization: British Columbia Cancer Agency (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NECTAR
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Prostate Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PAE (Experimental): Neoadjuvant PAE before RT
  Interventions: Procedure: Prostatic Artery Embolization

INTERVENTIONS:
Procedure: Prostatic Artery Embolization — PAE is a minimally invasive procedure that involves embolizing the arteries supplying the prostate, leading to its shrinkage.

SUMMARY:
The goal of this clinical trial is to find out whether prostate artery embolization (PAE) can help prevent or lessen urinary side effects caused by radiotherapy (RT) in people with prostate cancer, especially those who have larger prostates or urinary symptoms before treatment.

The main questions this study aims to answer are:

* Does PAE before RT reduce the severity of urinary side effects from RT?
* Does PAE affect the rates of genitourinary (GU) or gastrointestinal (GI) side effects after RT?

Researchers will look at changes in urinary symptoms from the start of the study to 6 months after PAE. They will also record any GU or GI side effects related to RT.

Participants will receive prostate artery embolization before starting radiotherapy, and complete questionnaires and assessments about GU and GI functions before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma with planned RT to the prostate
* Baseline (pre-PAE) prostate volume ≥ 50 cc
* Baseline (pre-PAE) IPSS ≥ 15
* If planned or ongoing ADT and/or 5-alpha reductase inhibitor (5ARI), patient should be on therapy for at least 12 weeks, and meet prostate volume and pre-PAE IPSS criteria at the time of enrollment.

Exclusion Criteria:

* Baseline (pre-PAE) IPSS storage/voiding ratio ≥ 1
* Previous prostate treatment (TURP, Laser therapies, MISTs)
* Chronic urinary retention requiring use of indwelling urinary catheter.
* Neurogenic bladder or other neurological disorder that is impacting bladder function (e.g., multiple sclerosis, Parkinson's disease, spinal cord injuries, etc.).
* Active urinary tract infections or recurrent urinary tract infections (>2/year), prostatitis, or interstitial cystitis.
* Receipt of beta blockers, antihistamines, anticonvulsants, or antispasmodics within 1 week of study treatment AND patient has not been on the same drug dosage for 6 months with a stable voiding pattern.
* Hypersensitivity reactions to contrast material not manageable with prophylaxis.
* Glomerular filtration rates less than 40 mL/min (unless on dialysis).
* Bilateral internal iliac arterial occlusion.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in LUTS symptoms measured by the IPSS at 6 months post-PAE | From enrollment to the 12 months after PAE

SECONDARY OUTCOMES:
Rates of Grade ≥2 GU and GI RT toxicity as assessed by CTCAE v5.0 | From enrollment to 12 months after PAE
Rates of PAE intraoperative and postoperative adverse events as assessed by Clavien-Dindo and CTCAE v5.0 | From the start of PAE to 12 months after PAE
Prostatic Specific antigen (PSA) at 6 months post-PAE | From enrollment to 12 months after PAE
Change in prostate volume calculated by TRUS at 6 months post-PAE | From enrollment to 12 months after PAE
Change in peak urinary flow rate (Qmax, ml/s) at 6 months post-PAE | From enrollment to 6 months after PAE
Change in postvoid residual urine (PVR, ml) at 6 months post-PAE | From enrollment to 6 months after PAE
Change in bladder and rectum mean RT dose from pre-PAE to pre-RT simulation scan | From pre-PAE simulation scan to pre-RT simulation scan
Urinary quality of life assessed by IPSS QoL scores | From enrollment to 12 months after PAE
Rate of local re-intervention for LUTS | From enrollment to 6 months after PAE
Erectile dysfunction assessed by the International Index of Erectile Function (IIEF-5) questionnaire | From enrollment to 12 months after PAE